CLINICAL TRIAL: NCT01563380
Title: Efficacy of Autologous Platelet Rich Plasma on Blood Loss, Pain, Wound Healing and Functional Outcome After Total Knee Arthroplasty by a Single Surgeon A Randomized, Prospective, Controlled, Double-blinded Study
Brief Title: Role of Autologous Platelet Rich Plasma in Total Knee Arthroplasty
Acronym: PRPTKA2012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Aditya K Aggarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: adi_agg_tka_prp-2012
Record Dates: First submitted 2012-03-15; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Blood Loss; Pain
Keywords: total knee arthroplasty; osteoarthritis; autologous Platelet rich plasma; complications; blood loss; Pain; functional outcome
MeSH Terms: conditions — Hemorrhage; Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP arm (Experimental): Platelet-rich plasma was applied over the wound including the capsule, medial and lateral recesses.
  Interventions: Biological: Platelet rich plasma
- Control Arm (No Intervention)

INTERVENTIONS:
Biological: Platelet rich plasma — PRP ready to be injected was supplied in a syringe in a quantity of 8 ml for each knee. The entire procedure was done under complete aseptic precautions. The calcium chloride required for activation was given in a separate syringe in a ratio of 4:1. About 12-16 ml of platelet rich plasma was obtained by this method and it was used for application. To confirm sterility, culture and sensitivity of PRP was performed. Patient's peripheral blood platelet count and the prepared platelet concentrate's platelet count was performed and recorded. Number of tramadol injections given was also noted
  Other Names: PRP; APG
  Arms: PRP arm

SUMMARY:
This study was designed to evaluate the efficacy of leucocyte free autologous platelet rich plasma on blood loss, pain, wound healing and functional outcome after total knee arthroplasty. The investigators hypothesized that application of platelet rich plasma would help in reducing blood loss, postoperative pain and expedite wound healing and better short-term functional outcome following total knee arthroplasty.

DETAILED DESCRIPTION:
Age, sex and BMI-matched patients who had unilateral or bilateral arthritis of the knee with similar deformity and preoperative range of motion were enrolled for this prospective randomized controlled double blinded clinical trial. The study was approved by the institutional review board, and all patients provided written informed consent to participate in it. Inclusion criteria were patient of either sex who underwent primary unilateral or bilateral surgery or the first surgery of a staged bilateral total knee replacement where the second stage was at least 6 weeks later and those who were willing and able to return for follow-up over at least a six month postoperative period. Patients with preoperative haemoglobin less than 10g/dl and with bleeding disorder were excluded from the study. Two Groups were assigned: 1) APG group and 2) Control group.

Demographic data of the patient was recorded. All routine investigations were carried out and the results were noted. Preoperative haemoglobin, range of motion, WOMAC8 scores and KSS9 scores were noted. Standard knee radiographs i.e. weight bearing anteroposterior and lateral views in 30 degree flexion were taken. Patients were randomly allocated to platelet gel group and control group using opaque envelope method which was opened on the day of surgery.

Pain was measured daily using VAS scale which consisted of markings from 1 to 10. Number of tramadol injections given was also noted. Hemoglobin was measured on the day of surgery and postop day 3 by sysmex automated analyser. Postoperative blood loss was also noted by measuring the weight of soaked dressing and converting it into blood volume. Number of blood units transfused was also recorded. Post operative wound dressing was done on day 3 except in case of soakage. Wound was assessed using wound score form. Similar physiotherapy was advised for both the groups. All the patients were advised isometric quadriceps and ankle pumping exercises on postoperative day 0 (POD0). Patients with less pain did the exercises on POD0 only. They were advocated range of motion exercises and straight leg raising on POD1. Patients with decreased pain and who were comfortable were ambulated with help of a walker on POD2. Range of motion was recorded on day 5, 6 weeks and 12 weeks and 6 months postoperatively. WOMAC scores and KSS scores were noted as shown in outcome evaluation.

Statistical analysis The statistical analysis was carried out using Statistical Package for Social Sciences (SPSS Inc., Chicago, IL, version 15.0 for Windows). All quantitative variables were estimated using measures of central location (mean, median) and measures of dispersion (standard deviation and standard error). Normality of data was checked by measures of skewness and Kolmogorov Smirnov tests of normality. For normally distributed data means were compared using student's t-test for two groups. For more than two groups ANOVA was applied. For Skewed data Mann-Whitney test was applied. Qualitative or categorical variables were described as frequencies and proportions. Proportions were compared using Chi square test. Sensitivity, specificity and diagnostic accuracy of different methods was calculated. All statistical tests were two-sided and were performed at a significance level of α=.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient of either sex who underwent primary unilateral or bilateral surgery or the first surgery of a staged bilateral total knee replacement where the second stage was at least 6 weeks later and those who were willing and able to return for follow-up over at least a six month postoperative period.

Exclusion Criteria:

* Patients with preoperative haemoglobin less than 10g/dl and with bleeding disorder were excluded from the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Total amount of Blood loss | participants will be followed on day of surgery, post op day 3
  Hemoglobin was measured on the day of surgery and postop day3 by sysmex automated analyser. Postoperative blood loss was also noted by measuring the weight of soaked dressing and converting it into blood volume. Number of blood units transfused was also recorded.

SECONDARY OUTCOMES:
Pain | participants will be followed upto an average of 12 weeks
  Pain was measured daily using VAS scale which consisted of markings from 1 to 10.
Wound healing | Participants will be followed upto an average of 3 weeks
  Wound was assessed using wound score form.
Range of motion | participants will be followed upto an average of 6months.
  Range of motion was recorded on day5, 6weeks and 12weeks and 6months postoperatively.
clinical outcome | Participants will be followed upto an average of 6months.
  Functional outcome was measured using both KSS and WOMAC scores. We assessed the patients at 6weeks, 12weeks and 6months.

CONTACTS AND LOCATIONS:
Overall Officials: Aditya K Aggarwal, MS DNB D Ort, Principal Investigator — Post graduate Institute of Medical Education & Research
Locations (1):
- Post graduate institute of Medical Education & Research, Chandigarh, Chandigarh, India